CLINICAL TRIAL: NCT04325893
Title: Hydroxychloroquine Versus Placebo in Patients Presenting COVID-19 Infection and at Risk of Secondary Complication: a Prospective, Multicentre, Randomised, Double-blind Study
Brief Title: Hydroxychloroquine Versus Placebo in COVID-19 Patients at Risk for Severe Disease
Acronym: HYCOVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: decrease in number of eligible patients
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49RC20_0071
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Active Comparator)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — First dose of 400 mg will be taken immediately after inclusion at day 0, the second dose of 400 mg will be taken on the same evening and at least 4 hours after the first dose. The treatment will then be continued for the following eight days at a rate of 200 mg in the morning and evening.
  Arms: Hydroxychloroquine
Drug: Placebo — TFirst dose of 400 mg will be taken immediately after inclusion at day 0, the second dose of 400 mg will be taken on the same evening and at least 4 hours after the first dose. The treatment will then be continued for the following eight days at a rate of 200 mg in the morning and evening.
  Arms: Placebo

SUMMARY:
A new human coronavirus responsible for pneumonia, SARS-CoV-2, emerged in China in December 2019 and has spread rapidly. COVID-19, the disease caused by this virus, has a very polymorphous clinical presentation, which ranges from upper respiratory tract infections to acute respiratory distress syndrome. It may appear serious straightaway or may evolve in two stages, with a worsening 7 to 10 days after the first clinical signs, potentially linked to a cytokine storm and accompanied by a high risk of thrombosis. The global mortality rate of COVID-19 is between 3% and 4%, with severe forms being more frequent among older patients. Management is symptomatic as no antiviral treatment has demonstrated any clinical benefit in this condition. Hydroxychloroquine is a derivative of chloroquine commonly used in some autoimmune diseases, such as systemic lupus erythematosus. It is active in vitro in cellular models of infection by many viruses such as HIV, hepatitis C or SARS-CoV. However, its interest in viral infections in humans has not been demonstrated.

Very recently, a preliminary uncontrolled study evaluated the effect of hydroxychloroquine on viral shedding in subjects with COVID-19. Among 20 patients treated with hydroxychloroquine at a dose of 600 mg per day, the percentage of patients with detectable SARS-CoV-2 RNA in the nasopharynx decreased from 100% at inclusion (start of treatment) to 43% six days later. In comparison, 15 of 16 untreated patients had a positive RT-PCR six days after inclusion. Furthermore, hydroxychloroquine has immunomodulating and anti-inflammatory properties, which could theoretically prevent or limit secondary worsening.

The research hypothesis is that treatment with hydroxychloroquine improves prognosis and reduces the risk of death or use for invasive ventilation in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Symptomatic infection with COVID-19 confirmed by positive RT-PCR SARS-CoV-2 or, failing that, by thorax CT-scan suggesting viral pneumopathy of peripheral predominance in a clinically significant context.
* Diagnosis in the previous two calendar days or, for an asymptomatic patient at the time of virological diagnosis, onset of symptoms in the previous two calendar days.
* Patient having at least one of the following risk factors for developing complications:

  * Age ≥75 years old
  * Age between 60 and 74 years old and presence of at least one comorbidity among the following: obesity (body mass index ≥ 30 kg/m²), arterial hypertension requiring treatment, diabetes mellitus requiring treatment
  * Need for supplemental oxygen to reach a peripheral capillary oxygen saturation of more than 94% (SpO2 > 94%), or a ratio of partial oxygen pressure to the fraction of inspired oxygen less than or equal to 300 mmHg (PaO2/FiO2 ≤ 300 mmHg).
* Patient affiliated to a social security scheme.
* Written and signed consent of the patient or a relative or emergency inclusion procedure.

Exclusion criteria

* Last RT-PCR negative for SARS-CoV-2
* Peripheral capillary oxygen saturation less than or equal to 94% (SpO2 ≤ 94%) despite oxygen therapy greater than or equal to 3 L/min (> 3 L/min)
* Organ failure requiring admission to a critical or intensive care unit.
* Comorbidity that is life threatening in the short-term (life expectancy < 3 months)
* Any reason that makes patient follow-up throughout the study impossible
* Current treatment with hydroxychloroquine
* Absolute contraindication to treatment with hydroxychloroquine (known hypersensitivity, retinopathy, concomitant treatment with risk of ventricular disorders, particularly torsades de pointe, known deficit of glucose-6-phosphate dehydrogenase, porphyria)
* Hypokalaemia < 3.5 mmol/L
* Corrected QT prolongation (QTc ≥ 440 ms in men and 460 ms in women).
* Child-Pugh's class C liver cirrhosis
* Chronic kidney failure with estimated GFR ≤ 30 ml/min, or ≤ 40 ml/min in patients with concomitant treatment with azithromycin
* Women who are pregnant, breastfeeding, or parturient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Number of death from any cause, or the need for intubation and mechanical ventilation during the 14 days following inclusion and start of treatment. | Day 14

SECONDARY OUTCOMES:
Number of death from any cause, or the need for intubation and mechanical ventilation during the 28 days following inclusion and start of treatment. | Day 28
Clinical evolution on the WHO Ordinal Scale for Clinical Improvement for COVID-19 between day 0 and day 14 | Day 14
  WHO Ordinal Scale for Clinical Improvement ranges from 0 to 8, higher score meaning poorer outcome
Clinical evolution on the WHO Ordinal Scale for Clinical Improvement for COVID-19 between day 0 and day 28. | Day 28
  WHO Ordinal Scale for Clinical Improvement ranges from 0 to 8, higher score meaning poorer outcome
Number of all-cause mortality at day 14 | Day 14
Number of all-cause mortality at day 28 | Day 28
Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal samples at day 5 | Day 5
Rate of positive SARS-CoV-2 RT-PCR on nasopharyngeal samples at day 10 | Day 10
The rate of venous thromboembolic events at day 28, documented and confirmed by an adjudication committee. | Day 28
Number of all-cause mortality at day 28 in patients aged 75 and older | day 28
Clinical evolution on the WHO OSCI scale for COVID-19 between day 0 and day 28 for patients aged 75 or older | day 28
Rate of severe adverse events at day 28 | day 28
Number of all-cause mortality at day 14 in patients aged 75 and older | day 14

CONTACTS AND LOCATIONS:
Locations (47):
- France (46):
  - CH Agen, Agen
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Auxerre, Auxerre
  - APHP Avicenne, Bobigny
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CH Chalon Sur Saône, Chalon-sur-Saône
  - CH Cherbroug, Cherbourg
  - CH Cholet, Cholet
  - CH Colmar, Colmar
  - CH Compiègne, Compiègne
  - APHP Henri Mondor, Créteil
  - CH Intercommunal Créteil, Créteil
  - CHU Dijon, Dijon
  - APHP Joffre Dupuytren, Draveil
  - CHD Vendée, La Roche-sur-Yon
  - CH Laval, Laval
  - CH Le Mans, Le Mans
  - CH Emile Roux, Le Puy-en-Velay
  - APHP Emile ROUX, Limeil-Brévannes
  - CHU Limoges, Limoges
  - CH Lorient, Lorient
  - Hôpital Européen - Marseille, Marseille
  - Hôpital Saint-Joseph, Marseille
  - CH Melun, Melun
  - CHU Nantes, Nantes
  - Hôpital Privé du Confluent, Nantes
  - CH Niort, Niort
  - CHR Orléans, Orléans
  - APHP Saint-Antoine, Paris
  - GH Croix Saint Simon, Paris
  - La Pitié-Salpétrière, Paris
  - CHU Poitiers, Poitiers
  - CH Pointoise, Pontoise
  - CH Quimper, Quimper
  - CH Saint-Brieuc, Saint-Brieuc
  - CHU Saint-Etienne, Saint-Etienne
  - CH Saint-Nazaire, Saint-Nazaire
  - CHU Toulouse, Toulouse
  - CH Tourcoing, Tourcoing
  - CHU Tours, Tours
  - CH Valenciennes, Valenciennes
  - Clinique Tessier Valenciennes, Valenciennes
  - CH Vannes, Vannes
  - CH Versailles, Versailles
- CH Princesse Grace, Monaco, Monaco

REFERENCES:
- [Derived] Dubee V, Roy PM, Vielle B, Parot-Schinkel E, Blanchet O, Darsonval A, Lefeuvre C, Abbara C, Boucher S, Devaud E, Robineau O, Rispal P, Guimard T, d'Anglejean E, Diamantis S, Custaud MA, Pellier I, Mercat A; HYCOVID study group; HYCOVID investigators; Angers University Hospital; Cholet Hospital; Laval Hospital; Le Mans Hospital; Tours University Hospital; Quimper Hospital; La Roche sur Yon Hospital; Tourcoing Hospital; Orleans Hospital; Nantes University Hospital; Niort Hospital; Lorient Hospital; Brest University Hospital; Cherbourg Hospital; Saint-Brieuc Hospital; Creteil - APHP University Hospital; Saint-Antoine - APHP University Hospital; Saint-Etienne University Hospital; Toulouse University Hospital; Melun Hospital; Dijon University Hospital; Princesse Grace - Monaco Hospital; Versailles Hospital; Colmar Hospital; Agen-Nerac Hospital; Caen University Hospital; Saint-Nazaire Hospital; Nantes - Confluent Hospital; Limoges University Hospital; Poitiers University Hospital; Amiens University Hospital; Bobigny - APHP University Hospital; Cergy-Pontoise Hospital; Valencienne Hospital; Valencienne - Clinique Tessier Hospital; Henri-Mondor - APHP University Hospital; Chalon-sur-Saone Hospital; Marseille European Hospital; Auxerre Hospital; Diaconnesses Croix-Saint-Simon Hospital; Marseille - Saint Joseph Hospital; HYCOVID management team: Steering committee (authors); HYCOVID management team: Independant data safety and monitoring board; HYCOVID management team: Independent adjudication of clinical events committee; Study management: Coordination; Study management: Data management. Hydroxychloroquine in mild-to-moderate coronavirus disease 2019: a placebo-controlled double blind trial. Clin Microbiol Infect. 2021 Aug;27(8):1124-1130. doi: 10.1016/j.cmi.2021.03.005. Epub 2021 Apr 1. PMID 33813110